CLINICAL TRIAL: NCT00616174
Title: The Effect of Maternal Warming During Cesarean Delivery on Neonatal Temperature
Brief Title: Does Warming Mothers During Cesarean Delivery Help Keep Babies Warm When Delivered?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H07-01490; H07-01490
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Cesarean Delivery
Keywords: Cesarean delivery; Active Warming; Neonatal Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Active warming with Bair Hugger blanket
  Interventions: Procedure: Active warming with Bair Hugger blanket

INTERVENTIONS:
Procedure: Active warming with Bair Hugger blanket — Standard care at BC Women's Hospital plus a Bair Hugger full access underbody blanket model 635 (Health Canada Licence # 12692) warmed by Bair Hugger temperature management unit model 750. Patient will lie on the underbody blanket and it will be turned on once patient is supine on operating table following the insertion of anesthetic. The warming device will be set to the medium temperature setting (380C). Warming will continue until the end of surgery unless otherwise requested by the mother.

SUMMARY:
The purpose of this study to investigate whether using a special warming blanket during Cesarean delivery helps maintain a normal body temperature in the baby when compared to mothers that are not warmed (standard care at BC Women's Hospital). Doctors observed that some babies have low body temperatures when they are born by Cesarean delivery. Since baby temperatures are dependant on the temperatures of their mothers, we believe that keeping the mother warm during surgery with the use of a special warming blanket that is filled with warm air will result in the baby being warmer at birth.

DETAILED DESCRIPTION:
Maternal hypothermia during Cesarean delivery is predominately caused by a combination of neuraxial anesthesia and exposure of abdominal contents and skin to the low temperatures of the operating room (OR). Since maternal temperature and fetal temperature are intimately related, neonates experience hypothermia at birth due to maternal hypothermia. Neonatal hypothermia on admission to the Intensive Care Unit is an important determinant of morbidity and mortality, particularly in preterm neonates.

At BC Women's Hospital the majority of Cesarean deliveries are done under neuraxial anesthesia and the pediatricians have observed that some babies had suboptimal body temperatures at the time of Cesarean delivery. The pediatricians wanted to reverse this trend in neonatal hypothermia and requested that the OR temperature be increased to 25oC, more in line with World Health Organization (WHO) guidelines for delivery rooms. However, raising OR temperatures is usually not a comfortable option to the majority of staff working in this environment, therefore WHO recommendations are not followed.

Forced air warming is a common technique used during surgical procedures to maintain normothermia in anesthetized patients. A bi-layered blanket with multiple air channels is connected to a warming device that forces warm air between the layers of the blanket and ultimately around the patient. This device is effective in warming hypothermic patients or maintaining temperature in normothermic patients in a cool OR.

The studies on maternal warming at Cesarean delivery that have been published to date have shown inconsistent findings thus the subject warrants further investigation.

We postulate that actively warming mothers will prevent or decrease the risk of neonatal hypothermia at birth. In addition, we will examine whether active warming has a larger effect in the premature neonate.

Neonatal axillary temperature at delivery will be our primary outcome.

Important variables measured include: neonatal umbilical vein pH, Apgar scores, maternal temperature throughout surgery (uterine incision -delivery time), presence of maternal shivering and maternal thermal comfort score.

This study will be a non-blinded, randomized controlled trial involving two groups:

1. Control group: Standard care i.e. cupboard warmed cotton blanket and cupboard warmed IV fluids.
2. Intervention group: Standard care as in control group plus a Bair Hugger full access underbody blanket model 635 (Health Canada Licence # 12692) warmed by Bair Hugger temperature management unit model 750. Patient will lie on the underbody blanket and it will be turned on once patient is supine on operating table following the insertion of anesthetic. The warming device will be set to the medium temperature setting (380C).

The intervention group will receive a forced air warming blanket throughout surgery.

The study will be conducted in the operating room at the BC Women's Hospital.

The target population is consenting, pregnant women undergoing either elective or urgent (no immediate threat to maternal or neonatal life but requiring delivery) Cesarean delivery under spinal or combined spinal-epidural anesthesia.

Exclusion factors include: emergency Cesarean deliveries or Cesarean deliveries under general anesthesia, mothers in active labor, mothers under 19 years old, those who cannot understand English, and lack of consent. Mothers with a suspected infection, Type I Diabetes Mellitus, a history of malignant hyperthermia and any disease/disorder that is known to affect temperature regulation will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing elective cesarean delivery under spinal anesthesia or combined spinal epidural anesthesia
* Greater than 28 weeks gestation
* ASA 1 & 2 classification of health
* Mothers presenting to the assessment or labour and delivery unit with ruptured membranes or early signs of labour, but not in active labour, who are not planned for a vaginal birth and who need an urgent cesarean delivery
* Potential subjects need to be able to read and understand English unless independent (non-partner) translator available

Exclusion Criteria:

* Mothers in active labour - 3cm or more dilated with regular coordinated contractions
* ASA 3 or above
* Emergency cesarean delivery for fetal heart rate abnormalities
* Cesarean delivery under general anesthesia
* Maternal age <19 years
* Maternal infection
* Mothers with a CSE where > 5ml of epidural local anesthetic is given prior to the delivery of the fetus
* Mothers with vascular disease - with the exception of hypertension/pre-eclampsia
* Mothers with Type I Diabetes Mellitus
* Untreated hypothyroidism or hyperthyroidism
* Mothers with a history or family history of malignant hyperthermia
* Those who cannot understand English, and lack of consent

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Neonatal axillary temperature at delivery | During delivery

CONTACTS AND LOCATIONS:
Overall Officials: Preston Roanne, MD, Principal Investigator — University of British Columbia; Joanne Douglas, MD, FRCPC, Study Director — University of British Columbia; Jason Reidy, MBBS, FRCA, Study Director — University of British Columbia; Simon Massey, MB BCh, MRCP, FRCA, Study Director — University of British Columbia; Rebecca Sherlock, MD, FRCPC, FAAP, PhD, Study Director — University of British Columbia; Jessica Tyler, BSc, Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada